CLINICAL TRIAL: NCT03201796
Title: Evaluation of the Efficacy and Safety of Prulifloxacin vs Levofloxacin in the Treatment of Chronic Bacterial Prostatitis.
Brief Title: Prulifloxacin in Chronic Bacterial Prostatitis (CBP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Hippocrates Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 027IC13250; 2014-003757-33 (EudraCT Number)
Record Dates: First submitted 2017-06-23; First posted 2017-06-28 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Chronic Bacterial Prostatitis
Keywords: Bacterial prostatitis; CBP; Levofloxacin; Prulifloxacin
MeSH Terms: conditions — Prostatitis | interventions — prulifloxacin; Levofloxacin

STUDY DESIGN:
Intervention Model Description: Double-blind, levofloxacin controlled, multicentre, international, prospective study.
Who Masked: Participant, Investigator
Masking Description: The present study will be performed in double blind condition. Consequently, during the study, neither the Investigator nor the patient will be aware of the treatment assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Prulifloxacin 600 mg
  Interventions: Drug: Prulifloxacin 600 mg
- Group 2 (Active Comparator): Levofloxacin 500 mg
  Interventions: Drug: Levofloxacin 500mg

INTERVENTIONS:
Drug: Prulifloxacin 600 mg — Oral administration of one tablet once daily for 28 days of prulifloxacin 600 mg. The investigational drug will be taken with a glass of water, preferably in the evening and at about the same time each day, 2 hours before or at least 4 hours after the eventual administration of cimetidine, antacids containing aluminum and magnesium or preparations containing iron and calcium.
  Other Names: Unidrox®
  Arms: Group 1
Drug: Levofloxacin 500mg — Oral administration of one tablet once daily for 28 days of levofloxacin 500 mg. The investigational drug will be taken with a glass of water, preferably in the evening and at about the same time each day, 2 hours before or at least 4 hours after the eventual administration of cimetidine, antacids containing aluminum and magnesium or preparations containing iron and calcium.
  Other Names: Levoxacin®
  Arms: Group 2

SUMMARY:
The aim of the study is to assess the efficacy and safety of prulifloxacin in comparison to levofloxacin in the treatment of patients affected by CBP.

DETAILED DESCRIPTION:
This is a randomized, double-blind, levofloxacin controlled, parallel group, multicentre, international, prospective study. The patients will be enrolled in the study and will be randomized to prulifloxacin or levofloxacin. Patient enrolment will be competitive.

The present study is planned to verify the microbiological and the clinical efficacy of a 28-day treatment period with prulifloxacin 600 mg in comparison with 28-day treatment period with levofloxacin 500 mg, both administered once daily, in patients with CBP. Safety and tolerability of a 28-day treatment period with prulifloxacin 600 mg will be also evaluated in comparison to levofloxacin 500 mg.

Levofloxacin 500 mg tablets has been selected as treatment comparator because it represents the drug of choice authorised for the treatment of CBP. Consequently, the dosage regimen to be administered to the patients is consistent with that reported in the relevant SPC.

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18 and 50 years of age (limited included) with no limitation of race.
2. Patients presenting symptoms of prostatitis for at least 3 months.
3. Laboratory evidence of CBP at Visit 0 (Screening), assessed by

   Meares&Stamey fourglass test and defined as:
   1. VB3 or EPS specimen containing ≥10^2 colony-forming units/ml of pathogen/s if the VB2 specimen is sterile; or
   2. VB3 or EPS specimen containing ≥10^2 colony-forming units/ml of pathogen/s different from any present in the VB2.
4. Medications for chronic prostatitis and/or medications that may affect bladder or prostate function (including but not limited to hormone therapy, anticholinergic or alpha blocker) must be discontinued at least 7 days before study drug intake.
5. Patients legally capable to give their consent to participate the study, and available to sign and date the written informed consent.

Exclusion Criteria:

1. Known hypersensitivity or allergy to antibacterial fluoroquinolones or to any components of the study medications.
2. Pathogen/s resistant to the study drugs at Visit 0 (Screening).
3. Suspicion for prostatic cancer, neurogenic bladder, Benign Prostatic Hypertrophy (BPH), bladder neck obstruction or urethral stricture.
4. Body Mass Index (BMI) < 16 kg/m^2.
5. Immunocompromised patients.
6. Signs or symptoms or clinical documentation for concurrent infections (including but not limited to sexually transmitted infections) and/or neoplasm.
7. Clinically significant abnormalities on physical examination, vital signs, ECG, laboratory tests at Visit 0 (Screening Visit).
8. Significant liver disease, defined as known active hepatitis or elevated liver enzymes > 3 times the upper boundary of the normal ranges.
9. Value of creatinine outside the normal ranges and judged clinically relevant by Investigator.
10. History of cardiac disease, including but not limited to myocardial infarction, heart failure, cardiomyopathy, cardiac hypertrophy, cardiac arrhythmias, bradycardia, cardiac conduction abnormalities, long QT syndrome.
11. Value of electrolytes (sodium, potassium, calcium, magnesium, chloride) outside the normal ranges and judged clinically relevant by Investigator.
12. Patients under treatment with medications that may cause increase of the QT interval.
13. History of tendinopathy.
14. Patients with latent or known deficiencies for the glucose-6-phosphate dehydrogenase, or with hereditary problems of galactose intolerance or the Lapp lactase deficiency or glucose-galactose malabsorption.
15. Recent or past history of psychiatric illness or epilepsy.
16. Treatment with antibiotics or antibacterials within 2 weeks before study drug start intake.
17. Treatment with experimental drugs (prulifloxacin or levofloxacin) or other fluoroquinolones within 4 weeks before study drug start intake.
18. Diabetic patients in treatment with oral hypoglycemic drugs and insulin.
19. Patients under treatment with corticosteroids or Non-Steroidal Antiflammatory Drugs (NSAIDs).
20. Concomitant treatment with xanthines or anticoagulant drugs or drugs producing hypokalemia or diuretics.
21. Positive history for drugs and alcohol abuse.
22. Inability to comply with the protocol requirements, instructions or study-related restrictions (i.e. uncooperative attitude, inability to return for study-visits, improbability of completing the clinical study).
23. Vulnerable subjects (i.e. persons kept in detention).
24. Subject involved in the conduct of the study (i.e. Investigator or his/her deputy, first grade relatives, pharmacist, assistant or other personnel).
25. Participation to an interventional clinical trial within 3 months prior to Visit 0 (Screening Visit).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 168 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Eradication of bacterial growth | 7 days after the EOT
  Eradication defined as absence of bacterial growth as <10^2 CFU/ml in voided bladder 3 (VB3) or expressed prostatic secretion (EPS) after 7 days from the End Of Treatment (EOT).

SECONDARY OUTCOMES:
Eradication of bacterial growth | 3 months after the EOT
  Eradication defined as absence of bacterial growth as <10^2 CFU/ml in voided bladder 3 (VB3) or expressed prostatic secretion (EPS) after 3 months from the EOT.
Eradication of bacterial growth | 6 months after the EOT
  Eradication defined as absence of bacterial growth as <10^2 CFU/ml in voided bladder 3 (VB3) or expressed prostatic secretion (EPS) after 6 months from the EOT.
Reduction in National Institute of Health - Chronic Prostatitis Symptom (NIH-CPSI) | Screening - 7 days after the EOT
  Reduction of total score in NIH-CPSI after 7 days from the EOT in comparison to the screening.
Reduction in National Institute of Health - Chronic Prostatitis Symptom (NIH-CPSI) | Screening - 3 months after the EOT
  Reduction of total score in NIH-CPSI after 3 months from the EOT in comparison to the screening.
Reduction in National Institute of Health - Chronic Prostatitis Symptom (NIH-CPSI) | Screening - 6 months after the EOT
  Reduction of total score in NIH-CPSI after 6 months from the EOT in comparison to the screening.
Frequency of treatment-related adverse events | 6 months
  Monitoring of the frequency of adverse events, physical examination, vital signs, ECG, laboratory analyses.

CONTACTS AND LOCATIONS:
Locations (11):
- Greece (2):
  - Urology Clinic General Hospital of Athens "GENNIMATAS", Athens
  - Urology Department General Hospital of Piraeus "TZANEIO", Piraeus
- Italy (9):
  - U.O. di Urologia- Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - U.O. Dipartimento della Donna, del bambino e delle malattie urologiche - Azienda ospedaliero- Universitaria e Policlinico di Bologna, Bologna
  - Urologia- Azienda Ospedaliero - Universitaria "Policlinico - Vittorio Emanuele", Catania
  - Clinica Urologica- Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - Azienda Ospedaliero-Universitaria "Careggi", Florence
  - Azienda Ospedaliera Universitaria "Federico II"- Dip. Di Ostreticia, ginecologia, Urologia, Napoli
  - Clinica Urologica del Dipartimento di Scienze Chirurgiche- Policlinico Universitario Agostino Gemelli di Roma, Roma
  - S.C. Urologia- AO "Città della Salute e della Scienza" di Torino - OSP.S. GIOV.BATTISTA MOLINETTE, Torino
  - Urologia- Ospedale di Trento- Presidio ospedaliero S. Chiara - Azienda Provinciale per i servizi sanitari (APSS), Trento

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.angelinipharma.com